CLINICAL TRIAL: NCT04576533
Title: Effects of Walking Out From Operating Room on Postoperative Recovery of Patients Undergoing Laparoscopic Colorectal Surgery
Brief Title: Patients Undergoing Laparoscopic Colorectal Surgery Walk Out From Operating Room After Surgery ( WOFOR-C1 )
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020ZSLYEC-137
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Enhanced Recovery After Surgery
Keywords: early mobilization

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- walk out from operating room (Experimental): patients will return to the ward after surgery by walking
  Interventions: Behavioral: walk out from operating room
- leave operating room by transporting bed (No Intervention): patients will return to the ward after surgery by lying on the transporting bed

INTERVENTIONS:
Behavioral: walk out from operating room — After the surgery of laparoscopic colectomy or laparoscopic rectectomy surgery (Dixon technique), patients will be encouraged to walk out from the operating room and return to the ward by walking under the condition of stable physiological parameters, painlessness, clear consciousness and normal muscle strength of lower limb
  Arms: walk out from operating room

SUMMARY:
Early mobilization is considered as an important strategy to enhance postoperative recovery. However, direct association between very early mobilization and improved recovery needs randomized control trials to prove. This study proposes the program of walking out from operating room (WOFOR) after surgery, which means that encouraging patients to walk out from the operating room and return to the ward by walking under the condition of painlessness, clear consciousness and normal muscle strength of lower limb. The aim of this randomized controlled trial is to investigate the effect of WOFOR on the postoperative recovery of patients undergoing laparoscopic colorectal surgery.

DETAILED DESCRIPTION:
Postoperative bed rest increases the risk of complications such as thromboembolism and intestinal adhesion. Encouraging early mobilization after surgery should be important, although actual effects of early mobilization still need randomized control trails to prove. The aim of this randomized controlled trial is to investigate the effect of walking out from operating room (very early mobilization after surgery) on the postoperative recovery of patients undergoing laparoscopic colorectal surgery.

A sample size of 300 patients in each group will be selected by a prior power analysis on the basis of the following assumptions: (1) an absolute reduction in the length of the hospital stay by 1 day ( 9 days in intervention group and 8 days in control group), (2) standard deviation 3 days, (3) α=0.05, (4) power 80% and .(5) missed follow-up rate 5%.

Patients will receive written and verbal information about the trial before written consent is obtained. The randomization will take place before the day of the surgery and the patients will be assigned to either intervention (return to ward by walking) or control group (return to ward by lying on the transporting bed ). A stratified randomization with three factors including sex(female or male), tumor site (colon or rectum) and age (18-40 or 41-65 years old ) will be performed to ensure an even spread. The randomization is performed using concealed allocation where envelopes are prepared externally using a randomization list prepared by a statistician.

The patients will receive general anesthesia combined with epidural analgesia. After surgery, the patients will be evaluated whether fulfilling the criteria for mobilization including stable physiological parameters, consciousness, normal level of orientation and muscle strength, and painlessness every ten minutes. If patients fulfill the criteria, they will receive different methods of returning to the ward based on the grouping. In the control group, the patient will return to the ward by lying on the transporting bed. In the intervention group, the patients will be raised to a sitting position for five minutes. If the patients do not complain any discomfort and have stable physiological parameters, they will be encouraged to stand. If standing do not cause any discomfort, they will be encouraged to walk within the range of 5-meter long and 60-centimeter wide. If patients can walk within the range, they will return to the surgical ward by walking under the protection of medical staffs.

Then, all study patients will be subject to the same management such as the guidance of drink and diet recovery, the guidance of mobilization in the ward (the duration and distance of walking in the ward will be recorded every day), nutrition supplement after surgery, and the criteria of drainage removal and hospital discharge. The outcomes such as the length of hospital stay after surgery will be recorded and analyzed to evaluate the effects of walking out from the operating room. The analysis of Intention-to-treat and Per-protocol-sets will be both performed by statisticians.

Summary statistics of mean (SD) for normally distributed data or median (IQR) for skewed data will be generated for continuous variables, and frequency (percentage) will be generated for categorical or ordinal variables. Continuous variables will be analyzed by Student's t test or Mann-Whitney U test or Repeated Measures Analysis of Variance, and categorical outcomes will be analyzed by χ² test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-65 Years old
* 2. scheduled for laparoscopic colectomy or laparoscopic rectectomy surgery (Dixon technique)
* 3. American Society of anesthesiology (ASA) grade I or grade II

Exclusion Criteria:

* 1. Patients have severe cardiac diseases (cardiac function grading greater than grade 3/arrhythmia including sick sinus syndrome, atrial fibrillation, atrial flutter, atrioventricular block, frequent ventricular premature, multiple ventricular premature, ventricular premature R on T, ventricular fibrillation and ventricular flutter/acute coronary syndrome) or respiratory failure or hepatic failure or renal failure;
* 2. Patients with poor blood glucose control (glycosylated hemoglobin>7%);
* 3. Patients with poor blood pressure control (receive regular antihypertensive medical treatment but still have systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg );
* 4. Patients have schizophrenia, epilepsy, Parkinson's disease, mental retardation, or hearing impairment.
* 5. Patients have thrombosis such as in lower extremity or in other veins.
* 6. Patients have neuromuscular disorders affecting lower limb activity, such as myasthenia gravis and cerebral infarction, which cause lower limb muscle weakness;
* 7. Patients have contraindications for epidural puncture.
* 8. Patients refuse to sign informed consent for research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay after surgery | at hospital discharge(expected 7 days after surgery)
  hospital stay time from operation completion to actual hospital discharge

SECONDARY OUTCOMES:
Time to fulfill the criteria of hospital discharge (recovery time) | expected 7 days after surgery
  The ideal time point for discharge, which is also considered as recovery time. The criteria for measuring recovery time included: 1) tolerance of diet and not necessary for intravenous nutrition; 2) analgesic-free, which is defined as visual analogue scale ≤3 without intravenous analgesic drugs, 3) adequate mobility; 4) afebrile status without major infectious complications
Re-admission incidence within 30 days after operation because of surgical complication | 30 days after operation
  Incidence of admit to hospital again within 30 days after operation because of surgical complication
Postoperative recovery score using 40-item quality of recovery scoring system(QoR-40) | at 1-day, 2-day, 3-day, 4-day after surgery and at hospital discharge (up to 8 days after surgery
  To evaluate the postoperative recovery using 40-item quality of recovery scoring system including emotional state (9items), physical comfort (12 items), physical independence (5 items), psychologic support (7 items), and pain (7 items).Each item is graded on a five-point Likert scale, and global scores range from 40 (extremely poor quality of recovery) to 200 (high quality of recovery)
Anxiety state evaluated by State-Trait Anxiety Inventory Form. The form used in this study is the Chinese version. | the day before surgery, and at 1-day, 2-day, 3-day, 4-day after surgery and at hospital discharge(up to 8 days after surgery
  The scales consist of 20 items; the responses range from 1 to 4 points (forced choice). The scores range from 20 (extremely low level of anxiety) to 80 (high level of anxiety). The State-Trait Anxiety Index classifies anxiety into five stages: stages 1 and 2 suggest mild anxiety; stage 3 suggests moderate anxiety, and stages 4 and 5 suggest severe anxiety
Severity of postoperative nausea and vomiting | at 1-day, 2-day after surgery(up to 2 days after surgery)
  Severity of postoperative nausea and vomiting is measured with the postoperative nausea and vomiting(PONV) intensity scale. Briefly, no PONV is defined as the absence of any emetic symptoms and nausea during the entire study period. Mild PONV is defined as the occurrence of mild nausea or one episode of vomiting if caused by an exogenous stimulus such as drinking or movement. Moderate PONV is reached when the patient vomits up to 2 times or experiences nausea that requires a rescue antiemetic therapy only once. Severe PONV is reached if the patient suffers more than two emetic episodes or needs more than one dose of a rescue antiemetic drugs.
Time to first flatus after surgery | at the time of first exhaust after surgery(expected average of 2 days after surgery)
  the time length between operation completion and the first flatus
Time to first defecation after surgery | at the time of the first defecation after surgery(expected average of 3 days after surgery)
  the time length between operation completion and the first defecation
The volume of drainage after surgery | expected average of 4 days after surgery
  Total volume of drainage after surgery and drainage volume at 24-hour and 48-hour after the end of surgery
Time to the removal of drainage tube | at the time of drainage removal(expected average of 4 days after surgery)
  recorded the time length between operation completion and the removal of drainage tube
Incidence of surgical complications within 30 days after surgery | 30 days after surgery
  Incidence of bleeding, wound infection, wound dehiscence within 30 days after surgery
Incidence of major cardiovascular and cerebrovascular adverse events within 30 days after operation | 30 days after surgery
  Incidence of a complex event consisting of all-cause death, myocardial infarction, stroke and emergency target vessel revascularization within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: SanQing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Chughtai B, Abraham C, Finn D, Rosenberg S, Yarlagadda B, Perrotti M. Fast track open partial nephrectomy: reduced postoperative length of stay with a goal-directed pathway does not compromise outcome. Adv Urol. 2008;2008:507543. doi: 10.1155/2008/507543. PMID 18784846
- [Background] Karl A, Buchner A, Becker A, Staehler M, Seitz M, Khoder W, Schneevoigt B, Weninger E, Rittler P, Grimm T, Gratzke C, Stief C. A new concept for early recovery after surgery for patients undergoing radical cystectomy for bladder cancer: results of a prospective randomized study. J Urol. 2014 Feb;191(2):335-40. doi: 10.1016/j.juro.2013.08.019. Epub 2013 Aug 19. PMID 23968966
- [Background] Barreca M, Renzi C, Tankel J, Shalhoub J, Sengupta N. Is there a role for enhanced recovery after laparoscopic bariatric surgery? Preliminary results from a specialist obesity treatment center. Surg Obes Relat Dis. 2016 Jan;12(1):119-26. doi: 10.1016/j.soard.2015.03.008. Epub 2015 Mar 20. PMID 25892343
- [Background] Collins JW, Patel H, Adding C, Annerstedt M, Dasgupta P, Khan SM, Artibani W, Gaston R, Piechaud T, Catto JW, Koupparis A, Rowe E, Perry M, Issa R, McGrath J, Kelly J, Schumacher M, Wijburg C, Canda AE, Balbay MD, Decaestecker K, Schwentner C, Stenzl A, Edeling S, Pokupic S, Stockle M, Siemer S, Sanchez-Salas R, Cathelineau X, Weston R, Johnson M, D'Hondt F, Mottrie A, Hosseini A, Wiklund PN. Enhanced Recovery After Robot-assisted Radical Cystectomy: EAU Robotic Urology Section Scientific Working Group Consensus View. Eur Urol. 2016 Oct;70(4):649-660. doi: 10.1016/j.eururo.2016.05.020. Epub 2016 May 24. PMID 27234997
- [Background] Patel HR, Cerantola Y, Valerio M, Persson B, Jichlinski P, Ljungqvist O, Hubner M, Kassouf W, Muller S, Baldini G, Carli F, Naesheim T, Ytrebo L, Revhaug A, Lassen K, Knutsen T, Aarsaether E, Wiklund P, Catto JW. Enhanced recovery after surgery: are we ready, and can we afford not to implement these pathways for patients undergoing radical cystectomy? Eur Urol. 2014 Feb;65(2):263-6. doi: 10.1016/j.eururo.2013.10.011. Epub 2013 Oct 22. PMID 24183418
- [Background] Palumbo V, Giannarini G, Crestani A, Rossanese M, Calandriello M, Ficarra V. Enhanced Recovery After Surgery Pathway in Patients Undergoing Open Radical Cystectomy Is Safe and Accelerates Bowel Function Recovery. Urology. 2018 May;115:125-132. doi: 10.1016/j.urology.2018.01.043. Epub 2018 Feb 15. PMID 29454972
- [Background] Azhar RA, Bochner B, Catto J, Goh AC, Kelly J, Patel HD, Pruthi RS, Thalmann GN, Desai M. Enhanced Recovery after Urological Surgery: A Contemporary Systematic Review of Outcomes, Key Elements, and Research Needs. Eur Urol. 2016 Jul;70(1):176-187. doi: 10.1016/j.eururo.2016.02.051. Epub 2016 Mar 9. PMID 26970912
- [Background] Tyson MD, Chang SS. Enhanced Recovery Pathways Versus Standard Care After Cystectomy: A Meta-analysis of the Effect on Perioperative Outcomes. Eur Urol. 2016 Dec;70(6):995-1003. doi: 10.1016/j.eururo.2016.05.031. Epub 2016 Jun 11. PMID 27297680
- [Background] Cerantola Y, Valerio M, Persson B, Jichlinski P, Ljungqvist O, Hubner M, Kassouf W, Muller S, Baldini G, Carli F, Naesheimh T, Ytrebo L, Revhaug A, Lassen K, Knutsen T, Aarsether E, Wiklund P, Patel HR. Guidelines for perioperative care after radical cystectomy for bladder cancer: Enhanced Recovery After Surgery (ERAS((R))) society recommendations. Clin Nutr. 2013 Dec;32(6):879-87. doi: 10.1016/j.clnu.2013.09.014. Epub 2013 Oct 17. PMID 24189391
- [Background] Semerjian A, Milbar N, Kates M, Gorin MA, Patel HD, Chalfin HJ, Frank SM, Wu CL, Yang WW, Hobson D, Robertson L, Wick E, Schoenberg MP, Pierorazio PM, Johnson MH, Stimson CJ, Bivalacqua TJ. Hospital Charges and Length of Stay Following Radical Cystectomy in the Enhanced Recovery After Surgery Era. Urology. 2018 Jan;111:86-91. doi: 10.1016/j.urology.2017.09.010. Epub 2017 Oct 13. PMID 29032237
- [Background] Sugi M, Matsuda T, Yoshida T, Taniguchi H, Mishima T, Yanishi M, Komai Y, Yasuda K, Kinoshita H, Yoshida K, Watanabe M. Introduction of an Enhanced Recovery after Surgery Protocol for Robot-Assisted Laparoscopic Radical Prostatectomy. Urol Int. 2017;99(2):194-200. doi: 10.1159/000457805. Epub 2017 Feb 17. PMID 28222423
- [Background] Lee TG, Kang SB, Kim DW, Hong S, Heo SC, Park KJ. Comparison of early mobilization and diet rehabilitation program with conventional care after laparoscopic colon surgery: a prospective randomized controlled trial. Dis Colon Rectum. 2011 Jan;54(1):21-8. doi: 10.1007/DCR.0b013e3181fcdb3e. PMID 21160309
- [Background] van der Leeden M, Huijsmans R, Geleijn E, de Lange-de Klerk ES, Dekker J, Bonjer HJ, van der Peet DL. Early enforced mobilisation following surgery for gastrointestinal cancer: feasibility and outcomes. Physiotherapy. 2016 Mar;102(1):103-10. doi: 10.1016/j.physio.2015.03.3722. Epub 2015 May 7. PMID 26059985
- [Background] Ni CY, Wang ZH, Huang ZP, Zhou H, Fu LJ, Cai H, Huang XX, Yang Y, Li HF, Zhou WP. Early enforced mobilization after liver resection: A prospective randomized controlled trial. Int J Surg. 2018 Jun;54(Pt A):254-258. doi: 10.1016/j.ijsu.2018.04.060. Epub 2018 May 9. PMID 29753000
- [Background] da Costa Torres D, Dos Santos PM, Reis HJ, Paisani DM, Chiavegato LD. Effectiveness of an early mobilization program on functional capacity after coronary artery bypass surgery: A randomized controlled trial protocol. SAGE Open Med. 2016 Dec 14;4:2050312116682256. doi: 10.1177/2050312116682256. eCollection 2016. PMID 28348739